CLINICAL TRIAL: NCT01023438
Title: Strategies To Improve Appropriate Prescribing In Heart Failure Patients. Assessment of the Effectiveness of an Integrated Clinical Pathway Between Cardiology and Primary Care Physicians to Implement Pharmacological Treatment
Brief Title: Strategies to Improve Prescribing in Heart Failure Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Up to sponsor decision
Sponsor: Niguarda Hospital (Other)
Collaborators: National Centre for Disease Prevention and Control (Unknown); Associazione Nazionale Medici Cardiologi Ospedalieri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SMART SC
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Assisted uptitration (Experimental): Uptitration of recommended drugs by primary care physician with specialist support
  Interventions: Other: Strategy for assisted uptitration
- Usual care (Active Comparator): Usual communication strategy from cardiologist to primary care physician
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Strategy for assisted uptitration — Active specialist support (mail, phone) and educational material provided to assist primary care physicians in drug uptitration
  Arms: Assisted uptitration
Other: Usual care — Usual communication strategy from cardiologist to primary care physician: uptitration advised but no active support nor educational material provided
  Arms: Usual care

SUMMARY:
The purpose of the study is to assess whether primary care physicians may uptitrate recommended drug therapies in stable heart failure patients if educational material and specialist support including phone or mail consultation are provided

DETAILED DESCRIPTION:
Heart failure is highly prevalent, particularly in elderly subjects, and costly, mainly because of the high rate of recurrent hospital admissions. Although guideline-recommended treatments, such as beta-blockers and renin-angiotensin inhibitors, are effective on both mortality and morbidity, these drugs are very often underprescribed or used at lower doses than those shown to be beneficial in clinical trials, particularly in the primary care setting, for fear of adverse events. Although referral to specialist services may improve prescription of recommended drugs and doses achieved, frequent consultations may be unfeasible and costly.The study is designed to assess whether active specialist support and educational material improve the prescription process for heart failure patients in primary care

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of heart failure wih depressed systolic function (left ventricular ejection fraction <40% in the previous 6 months).
* stable NYHA class II-III
* a clinical indication to implement drug therapy with betablockers and/or renin-angiotensin system inhibitors and current dose <50% of the target dose

Exclusion Criteria:

* NYHA class IV or clinically unstable
* cardiac surgery or cardiac resynchronization therapy planned within the following 6 months
* discharged to a rehabilitation unit refusal or impossibility to present to outpatient visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
achievement of ≥ 50% of the target dose either for beta-blockers (12.5mg b.i.d. for carvedilol, 5mg u.i.d for bisoprolol) or for ACE-inhibitors or angiotensin-receptor blockers in patients in whom beta-blockers are contraindicated | 12 weeks

SECONDARY OUTCOMES:
achievement of ≥ 50% of the target dose of both beta-blockers and ACE-inhibitors or angiotensin-receptor blockers | 12 weeks
proportion of patients who started drug uptitration by week 12 expressed as N° patients in whom therapy was uptitrated by their primary care physician/N° randomized patients | 12 weeks
all cause death, hospital admissions, emergency room visits; changes in quality of life by SF12, a generic questionnaire | 12 weeks
value of DRG reimbursement for hospital admissions and specialist visits | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Di Lenarda, MD, Study Chair — Cardiovascular Center ASS 1 Triestina, Trieste Italy; Fabrizio Oliva, MD, Study Chair — Heart Failure Heart Transplant Program, Cardiovascular Department, Niguarda Hospital, Milan, Italy
Locations (1):
- Azienda Opsedaliera Ospedale Niguarda Ca' Granda, Milan, MI, Italy

REFERENCES:
- See also: official website of the Study Sponsor Italian Association of Hospital Cardiologists — http://www.anmco.it